CLINICAL TRIAL: NCT02466672
Title: The Role and Effect of Anemia in Children With Pneumonia
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Mbarara University of Science and Technology (Other); Thrasher Research Fund (Other); National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Peter Moschovis, Postdoctoral Fellow, Massachusetts General Hospital
Other Study IDs: 2014P001325; 5F32HL124951-03 (NIH)
Record Dates: First submitted 2015-06-03; First posted 2015-06-09 (Estimated); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Anemia; Pneumonia
MeSH Terms: conditions — Anemia; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: none - observational only

SUMMARY:
This study will measure the effect of anemia on the outcomes of hospitalized children with severe pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months to 59 months
* WHO-defined severe pneumonia

Exclusion Criteria:

* Congenital heart disease

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children age 6 months to 59 months admitted to the hospital with WHO-defined severe pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2015-02; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Time to recovery from pneumonia | participants will be followed for the duration of hospital stay, an expected average of 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Peter P Moschovis, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Mbarara University of Science and Technology, Mbarara, Uganda